CLINICAL TRIAL: NCT01901055
Title: The Effect of Treatment of Obstructive Sleep Apnea on Diabetes Self Management and Glycemic Control
Brief Title: Diabetes-Obstructive Sleep Apnea Treatment Trial
Acronym: DOTT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study did not reach 50% of the proposed sample size. Recruitment slow because persons not interested in being randomized to a sham-control CPAP device or not CPAP naïve.
Sponsor: Eileen R. Chasens (Other)
Responsible Party: Sponsor-Investigator, Eileen R. Chasens, Professor of Nursing, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 5R01DK096028-02 (NIH)
Record Dates: First submitted 2013-07-10; First posted 2013-07-17 (Estimated); Results first posted 2021-08-13 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-08

CONDITIONS: Type 2 Diabetes; Obstructive Sleep Apnea
Keywords: sleep apnea; diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Sleep Apnea, Obstructive; Sleep Apnea Syndromes; Diabetes Mellitus | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Intervention Model Description: Parallel was a one-way cross over after 12 weeks with persons originally in the sham group being titrated onto active CPAP.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active CPAP treatment (Experimental): Treatment of obstructive sleep apnea with continuous positive airway pressure (CPAP)
  Interventions: Device: CPAP; Behavioral: Diabetes Education
- Sham-CPAP (Placebo Comparator): Device that appears like the treatment of obstructive sleep apnea, a continuous positive airway pressure device, but that does not provide treatment.
  Interventions: Device: CPAP; Device: Sham-CPAP; Behavioral: Diabetes Education

INTERVENTIONS:
Device: CPAP — CPAP is a device that has a mask worn over the nose that is attached to a device that provides positive airway pressure. CPAP is worn while sleeping, it splints open the airway and prevent apneas (cessation of breathing) and hypopneas (reduced airflow while breathing).
  Other Names: Continuous Positive Airway Pressure
Device: Sham-CPAP — Sham-CPAP is a device that has a mask worn over the nose that is attached to a device that looks and sounds like CPAP however it does not provide positive airway pressure. Sham-CPAP is worn while sleeping, it does not splint open the airway and prevent apneas (cessation of breathing) and hypopneas (reduced airflow while breathing).
  Other Names: Sham Continuous Positive Airway Pressure
  Arms: Sham-CPAP
Behavioral: Diabetes Education — Diabetes Education will be delivered to participants in both the CPAP group and the Sham-CPAP group. The education will be based on ADA and AADE guidelines and consist of 2 in-person sessions (90 minutes and 60 minutes) and 3 follow-up phone calls 9about 15 minutes each)

SUMMARY:
Diabetes self-management is important to help adults with type 2 diabetes achieve glucose control. Obstructive sleep apnea often co-exists with type 2 diabetes and may act as a barrier to diabetes self-management and glucose control. We will examine if treatment of obstructive sleep apnea with continuous positive airway pressure (CPAP), combined with diabetes education, results in improved diabetes self-management and glucose control.

DETAILED DESCRIPTION:
While diabetes self-management has been improved and refined over the last 30 years, many persons with T2DM continue to have difficulty in achieving glycemic goals. Obstructive sleep apnea (OSA) has a high prevalence among adults with type 2 diabetes (T2DM) and is associated with excessive daytime sleepiness, impaired mood, decreased vigilance, and reduced functional outcomes. The degree that OSA affects diabetes self-management, a known determinant of glycemic control, remains unstudied.

The most effective treatment for OSA, continuous positive airway pressure (CPAP), results in improved self-reported daytime functioning. However, the effect of CPAP treatment on reception of diabetes education remains unknown. The underlying premise of the proposed study from this new investigator is that OSA hinders diabetes self-management in adults with T2DM.

Our goal is to improve understanding of the effect of OSA on diabetes self-management and to determine the efficacy of CPAP treatment in improving diabetes outcomes in adults treated with CPAP compared to those on sham-CPAP. Expanding our understanding of the effect of sleep disturbances on diabetes self-management may lead to improved guidelines for screening and treatment of OSA in the increasingly large portion of the population with diabetes

ELIGIBILITY:
Inclusion Criteria:

* Suboptimal glucose control (A1C ≥ 6.5%)
* Moderate-to-severe obstructive sleep apnea (apnea + hypopnea index >= 10/hour)
* age 18 years and older

Exclusion Criteria:

* Poor glucose control (A1C > 11)
* Type 1 or gestational diabetes
* Sleep duration < 4 hrs
* Acute medical or surgical conditions or hospitalization ≤ 3 months
* Oxygen or bi-level PAP required
* Prior CPAP or persons in household with CPAP
* Employed in safety sensitive job
* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2014-02-13 (Actual); Primary Completion 2019-05-08 (Actual); Study Completion 2019-05-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eileen R. Chasens, PhD, Principal Investigator — University of Pittsburgh
Locations (4):
- United States (4):
  - John D. Dingell VAMC, Detroit, Michigan
  - Pittsburgh Veterans Administration Medical Center, Pittsburgh, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - West Virginia University, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Imes CC, Bizhanova Z, Sereika SM, Korytkowski MT, Atwood CW Jr, Burke LE, Kariuki J, Morris JL, Stansbury R, Strollo PJ Jr, Chasens ER. Metabolic outcomes in adults with type 2 diabetes and sleep disorders. Sleep Breath. 2022 Mar;26(1):339-346. doi: 10.1007/s11325-021-02408-x. Epub 2021 Jun 9. PMID 34105104
- [Derived] Chasens ER, Atwood CW, Burke LE, Korytkowski M, Stansbury R, Strollo PJ, Sereika SM. Diabetes sleep treatment trial: Premise, design, and methodology. Contemp Clin Trials. 2019 Jan;76:104-111. doi: 10.1016/j.cct.2018.11.014. Epub 2018 Dec 2. PMID 30517889

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruitment started in 2014 and the last participant was evaluated in 2019. The total sample screened (N=862) was from the University of Pittsburgh (n=720), Veterans Administration Pittsburgh Healthcare System (n=58), West Virginial University (n=72), and the John Dingell Detroit Veterans Administration Healthcare System (n=12).
Pre-assignment Details: Phone assessment excluded persons with prior CPAP use, not having diagnosis of type 2 diabetes, history of a sleepiness related accident or near miss, or not ambulatory.
  Participants (n=355) who met the phone screening were invited for a baseline assessment. The baseline assessment excluded persons with HbA1c either < 6.5% or > 11%; without OSA, with too high a AHI or severe oxygen desaturations, or not interested in being randomized to sham-CPAP. 98 participants meet all eligibility criteria.
Period: Randomization But Not Titrated
Arm/Group | Active CPAP Treatment | Sham-CPAP
Started (49 Subjects were randomized to each group. Milestone is that they completed overnight sleep study and were successfully titrated to CPAP or sham-CPAP/) | 49 | 49
Completed | 48 | 47
Not Completed | 1 | 2
Not completed — Did not come to titration study | 1 | 1
Not completed — Physician Decision | 0 | 1
Period: Started Protocol to Week 6
Arm/Group | Active CPAP Treatment | Sham-CPAP
Started | 48 | 47
Completed | 45 | 43
Not Completed | 3 | 4
Not completed — Physician Decision | 2 | 1
Not completed — complains of difficulty with wearing mask | 0 | 2
Not completed — Participant had not disclosed that they had been previously been on CPAP | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1
Period: Week 12 Assessment
Arm/Group | Active CPAP Treatment | Sham-CPAP
Started | 45 | 43
Completed | 44 | 39
Not Completed | 1 | 4
Not completed — Medical procedure that may interfere with wearing CPAPP mask | 1 | 0
Not completed — Withdrawal by Subject | 0 | 4
Period: Week 24
Arm/Group | Active CPAP Treatment | Sham-CPAP
Started (This is the final assessment of persons on active CPAP treatment. After the 12 week assessment, all participant were told their group assignment. Those on sham-CPAP were allowed to titrate to active CPAP. This assessment (week 24 in protocol) is 12 weeks after the participants started active treatment.) | 44 | 39
Completed | 30 | 20
Not Completed | 14 | 19
Not completed — Withdrawal by Subject | 13 | 19
Not completed — Physician Decision | 1 | 0
Period: Week 36
Arm/Group | Active CPAP Treatment | Sham-CPAP
Started | 30 | 20
Completed (Only participants originally in the sham-CPAP group were in this time period where they completed being on 24 weeks active CPAP.) | 30 | 15
Not Completed | 0 | 5
Not completed — Withdrawal by Subject | 0 | 5

BASELINE CHARACTERISTICS:
Population: Participants who were initially approved by primary care provider to engage in study with type 2 diabetes, an HbA1c 6.5% to 11.0%, age 18 years or older, apnea-hypopnea index >= 10/hr., denied excessive alcohol consumption, denied car crash or near accident, denied previous CPAP use, denied being pregnant or negative test if potentially pregnant, and willing to be randomized to participate in study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Active CPAP Treatment | Sham-CPAP | Total
Number analyzed (Participants) | 49 | 49 | 98
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 31 | 38 | 69
  >=65 years | 18 | 11 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.08 (10.13) | 57.37 (9.32) | 58.72 (9.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 19 | 42
  Male | 26 | 30 | 56
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 48 | 48 | 96
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 8 | 21
  White | 36 | 37 | 73
  More than one race | 0 | 3 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 49 | 49 | 98
HbA1c [Mean (Standard Deviation); unit: percentage of glycated hemoglobins] — Percentage of the number of hemoglobin molecules on red blood cells that are glycated. HbA1c indicates overall glucose control over last 3 months. Reference range for adults without diabetes is 4-5.9%.
  percentage of glycated hemoglobins | 7.73 (0.75) | 8.04 (1.01) | 7.89 (0.90)
Fructosamine [Mean (Standard Deviation); unit: µmol/L] — Glucose molecules permanently combined with albumin proteins in the blood, fructosamine indicates the average level of blood glucose control over the past 2-3 weeks. Normal range in persons without diabetes is is 200-285 µmol/L. Population: This measure was not done by protocol at University of West Virginia and Detroit VA; missing data at Pitt and VAPHS
  µmol/L
    number analyzed (Participants) | 41 | 42 | 83
    (all) | 285.10 (45.20) | 301.88 (54.41) | 293.59 (50.48)
Body Mass Index (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] — Obtained by measured height and weight.
  kg/m^2 | 35.71 (6.16) | 36.69 (6.99) | 36.20 (6.57)
Apnea-Hypopnea Index [Mean (Standard Deviation); unit: events per hour of sleep] — Mean number of apneas (cessation of breathing) and hypopneas (reduction in airflow by at least 50%) during overnight home sleep study with portable device that measures nasal airflow, chest and abdominal movement, oximetry, EKG.
  events per hour of sleep | 22.48 (13.41) | 25.92 (15.86) | 24.20 (14.71)
Epworth Sleepiness Scale [Mean (Standard Deviation); unit: units on a scale] — Validated instrument to measure subjective sleepiness. Scores potentially range from 0 to 24 with higher scores indicating more sleepiness.
  units on a scale | 10.22 (4.36) | 10.39 (4.76) | 10.31 (4.54)
Pittsburgh Sleep Quality Index Total Score [Mean (Standard Deviation); unit: units on a scale] — The Pittsburgh Sleep Quality Index (PSQI) is a validated measure of dimensions of sleep quality. Higher scores indicate worse sleep quality; potential range is 0 to 27 with scores greater than 5 indicating poor sleep quality.
  units on a scale | 10.00 (3.61) | 9.67 (4.19) | 9.84 (3.89)

OUTCOME MEASURES:

1. Primary Outcome: HbA1C Level
Description: Glycated hemoglobin test that estimates the blood glucose level over last 2 to 3 months. Higher scores indicate worse diabetes control.
Time Frame: baseline, 6 weeks, 12 weeks
Population: All randomized participants were analyzed (the intention to treat method).
Measure: Mean (Standard Error); unit: % of glycated hemoglobin in the blood
Groups:
- Sham-CPAP Treatment: Device that appears like the treatment of obstructive sleep apnea, a continuous positive airway pressure device, but that does not provide treatment.
Arm/Group | Active CPAP Treatment | Sham-CPAP Treatment
Number analyzed (Participants) | 49 | 49
% of glycated hemoglobin in the blood
  Baseline | 7.73 (0.13) | 8.04 (0.13)
  6-week | 7.49 (0.17) | 820 (0.17)
  12-week | 7.46 (0.15) | 7.80 (0.16)
Statistical Analysis 1: Comparison: Active CPAP Treatment vs Sham-CPAP Treatment; Statistical analyses were revised from the original protocol for reporting results at 24 week because unable to recruit an adequate sample size at this time point of participants originally on CPAP for 24 weeks and those who were in the original sham-CPAP group who crossed over to CPAP and completed 24 weeks of treatment; Test type: Superiority; p = 0.017, Mixed Models Analysis — F-test statistics for group X time = 4.27; Mean Difference (Net) = -0.32, 95% CI 2-sided [-0.68 to 0.04], Standard Error of Mean 0.18 — Treatment Difference = Active CPAP - Sham CPAP

2. Secondary Outcome: Fructosamine Level
Description: Measurement of glucose in plasma that estimates the blood glucose level over last 10 days to 3 weeks. The normal range is from 221.00 to 451.00.
Time Frame: baseline, 6 weeks, 12 weeks
Population: All randomized participants with data were analyzed (the intention to treat method). Unable to obtain laboratory value on from participants from West Virginia University (n=12), Detroit (n=1), and Pitt (n=2)
Measure: Mean (Standard Error); unit: umol/L (micromols per liter)
Arm/Group | Active CPAP Treatment | Sham-CPAP
Number analyzed (Participants) | 41 | 42
umol/L (micromols per liter)
  Baseline | 285.94 (7.78) | 300.99 (7.68)
  6-week | 272.84 (7.32) | 293.73 (7.53)
  12-week | 274.87 (7.53) | 285.56 (7.80)
Statistical Analysis 1: Comparison: Active CPAP Treatment vs Sham-CPAP; Test type: Superiority; p = 0.307, Mixed Models Analysis — F test statistics for group X time = 1.20; Mean Difference (Net) = -16.78, 95% CI 2-sided [-38.66 to 5.09], Standard Error of Mean 10.99 — Treatment Difference = Active CPAP - Sham CPAP

3. Secondary Outcome: Diabetes Diet Adherence
Description: Diabetes Diet Adherence score from the Summary of Diabetes Self-Care Activities (SDSCA) Questionnaire, Average number of days each week that was adherent to diabetes diet, range from minimum=0 days to maximum=7 days; higher number indicates better adherence to diabetes diet
Time Frame: baseline, 6 weeks, 12 weeks
Population: All randomized participants with valid data were analyzed (the intention to treat method). One participant with missing data.
Measure: Mean (Standard Error); unit: Average number of days/week
Arm/Group | Active CPAP Treatment | Sham-CPAP
Number analyzed (Participants) | 49 | 48
Average number of days/week
  Baseline | 3.55 (0.29) | 3.61 (0.30)
  6-week | 4.18 (0.27) | 4.05 (0.29)
  12-week | 4.30 (0.25) | 4.05 (0.27)
Statistical Analysis 1: Comparison: Active CPAP Treatment vs Sham-CPAP; Test type: Superiority; p = 0.732, Mixed Models Analysis — F test statistics for group X time = 0.31; Mean Difference (Net) = -0.25, 95% CI 2-sided [-0.85 to 0.35], Standard Error of Mean 0.30 — Treatment Difference = Active CPAP - Sham CPAP

4. Secondary Outcome: Diabetes Knowledge
Description: Score on the Diabetes Knowledge Test. Scores range minimum=0 to maximum=100, higher scores indicate higher knowledge (this measure only done at 12 weeks)
Time Frame: baseline,12 weeks only
Population: All randomized participants were analyzed (the intention to treat method).
Measure: Mean (Standard Error); unit: % of correct answers
Arm/Group | Active CPAP Treatment | Sham-CPAP
Number analyzed (Participants) | 49 | 49
% of correct answers
  Baseline | 79.39 (1.88) | 75.74 (1.88)
  12-week | 83.20 (1.79) | 79.81 (1.88)
Statistical Analysis 1: Comparison: Active CPAP Treatment vs Sham-CPAP; Test type: Superiority; p = 0.919, Mixed Models Analysis — F test statistics for group X time = 0.01; Mean Difference (Net) = 3.65, 95% CI 2-sided [-1.62 to 8.92], Standard Error of Mean 2.65 — Treatment Difference = Active CPAP - Sham CPAP

5. Secondary Outcome: Self-Monitoring of Blood Glucose (SMBG)
Description: SMBG score from the Summary of Diabetes Self-Care Activities (SDSCA) Questionnaire, Average number of days each week that SMBG was done, range from 0 days to 7 days; higher number indicates better SMBG
Time Frame: baseline, 6 weeks, 12 weeks
Population: All randomized participants were analyzed (the intention to treat method).
Measure: Mean (Standard Error); unit: Average number of days/week
Arm/Group | Active CPAP Treatment | Sham-CPAP
Number analyzed (Participants) | 49 | 49
Average number of days/week
  Baseline: number analyzed (Participants) | 49 | 48
  Baseline | 4.17 (0.38) | 4.24 (0.38)
  6-week: number analyzed (Participants) | 49 | 48
  6-week | 5.44 (0.31) | 5.10 (0.33)
  12-week: number analyzed (Participants) | 49 | 48
  12-week | 5.52 (0.34) | 4.61 (0.36)
Statistical Analysis 1: Comparison: Active CPAP Treatment vs Sham-CPAP; Test type: Superiority; p = 0.125, Mixed Models Analysis — F-test statistics for group X time = 2.12; Mean Difference (Net) = -0.11, 95% CI 2-sided [-1.18 to 0.96], Standard Error of Mean 0.54 — Treatment Difference = Active CPAP - Sham CPAP

6. Secondary Outcome: Steps Walked
Description: Average number of steps walked daily; measured by BodyMedia Armband; higher numbers indicate more steps walked. The range is from 397.83 to 16839.00.
Time Frame: baseline, 6 weeks, 12 weeks
Population: All randomized participants were analyzed (the intention to treat method).
Measure: Mean (Standard Error); unit: Steps/day
Arm/Group | Active CPAP Treatment | Sham-CPAP
Number analyzed (Participants) | 49 | 49
Steps/day
  Baseline | 4550.83 (374.15) | 4463.61 (374.15)
  6-week | 4774.81 (386.56) | 4240.42 (403.84)
  12-week | 4741.43 (355.27) | 4403.97 (372.96)
Statistical Analysis 1: Comparison: Active CPAP Treatment vs Sham-CPAP; Test type: Superiority; p = 0.639, Mixed Models Analysis — F-test statistics for group X time = 0.45; Mean Difference (Net) = 87.22, 95% CI 2-sided [-936.10 to 1137.50], Standard Error of Mean 529.10 — Treatment Difference = Active CPAP - Sham CPAP

7. Secondary Outcome: Self-Monitoring of Foot Care
Description: Foot Care score from the Summary of Diabetes Self-Care Activities (SDSCA) Questionnaire, Average number of days each week that foot care was done, range from 0 days to 7 days; higher number indicates better adherence to foot care
Time Frame: baseline, 6 weeks, 12 weeks
Population: All randomized participants were analyzed (the intention to treat method).
Measure: Mean (Standard Error); unit: Average number of days/week
Arm/Group | Active CPAP Treatment | Sham-CPAP
Number analyzed (Participants) | 49 | 49
Average number of days/week
  Baseline: number analyzed (Participants) | 49 | 48
  Baseline | 3.26 (0.35) | 3.89 (0.35)
  6-week: number analyzed (Participants) | 49 | 48
  6-week | 3.56 (0.37) | 4.44 (0.39)
  12-week: number analyzed (Participants) | 49 | 48
  12-week | 4.18 (0.37) | 4.57 (0.39)
Statistical Analysis 1: Comparison: Active CPAP Treatment vs Sham-CPAP; Test type: Superiority; p = 0.461, Mixed Models Analysis — F-test statistics for group X time = 0.78; Mean Difference (Net) = -0.63, 95% CI 2-sided [-1.61 to 0.35], Standard Error of Mean 0.49 — Treatment Difference = Active CPAP - Sham CPAP

8. Secondary Outcome: Diabetes-Related Distress
Description: Score of the Problem Areas in Diabetes (PAID) Questionnaire; scores range from 0-100, higher scores indicate worse diabetes-related distress.
Time Frame: baseline, 6 weeks, 12 weeks
Population: All randomized participants were analyzed (the intention to treat method).
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Active CPAP Treatment | Sham-CPAP
Number analyzed (Participants) | 49 | 49
score on a scale
  Baseline: number analyzed (Participants) | 49 | 48
  Baseline | 29.18 (2.77) | 26.44 (2.79)
  6-week: number analyzed (Participants) | 49 | 48
  6-week | 22.75 (2.72) | 20.08 (2.81)
  12-week: number analyzed (Participants) | 49 | 48
  12-week | 20.7413 (2.60) | 19.99 (2.76)
Statistical Analysis 1: Comparison: Active CPAP Treatment vs Sham-CPAP; Test type: Superiority; p = 0.776, Mixed Models Analysis — F-test statistics for group X time= 0.25; Mean Difference (Net) = 3.04, 95% CI 2-sided [-4.78 to 10.86], Standard Error of Mean 3.94 — Treatment Difference = Active CPAP - Sham CPAP

9. Secondary Outcome: Sleep Quality
Description: Sleep Quality is measured by the Pittsburgh Sleep Quality Index (PSQI) - Higher scores indicate worse sleep quality. The potential range is from 0 to 27 with higher scores indicating worse sleep quality.
Time Frame: baseline, 6 weeks, 12 weeks
Population: All randomized participants were analyzed (the intention to treat method).
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Active CPAP Treatment | Sham-CPAP
Number analyzed (Participants) | 49 | 49
score on a scale
  Baseline | 10.00 (0.56) | 9.67 (0.56)
  6-week | 8.12 (0.52) | 8.57 (0.54)
  12-week | 8.77 (0.55) | 8.54 (0.59)
Statistical Analysis 1: Comparison: Active CPAP Treatment vs Sham-CPAP; Test type: Superiority; p = 0.378, Mixed Models Analysis — F-test statistics for group X time = 0.98; Mean Difference (Net) = 0.33, 95% CI 2-sided [-1.24 to 1.89], Standard Error of Mean 0.79 — Treatment Difference = Active CPAP - Sham CPAP

10. Secondary Outcome: Mood
Description: Mood impairment measured by the Profile of Mood States (POMS) total score; potential scores range from 0 to 60; higher scores indicate worse mood.
Time Frame: baseline, 6 weeks, 12 weeks
Population: All randomized participants were analyzed (the intention to treat method).
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Active CPAP Treatment | Sham-CPAP Treatment
Number analyzed (Participants) | 49 | 49
score on a scale
  Baseline | 28.94 (5.12) | 25.76 (5.12)
  6-week | 17.28 (5.35) | 23.17 (5.49)
  12-week | 19.32 (5.85) | 22.61 (6.10)
Statistical Analysis 1: Comparison: Active CPAP Treatment vs Sham-CPAP Treatment; Test type: Superiority; p = 0.213, Mixed Models Analysis — F-test statistics for group X time = 1.57; Mean Difference (Net) = 3.18, 95% CI 2-sided [-11.19 to 17.56], Standard Error of Mean 7.24 — Treatment Difference = Active CPAP - Sham CPAP

11. Secondary Outcome: Vigilance
Description: Ability to maintain attention (i.e. vigilance); Measured by the Psychomotor Vigilance Test primary metric being transformed lapses (i.e. when person does not respond to a visual stimuli in a reaction time test). Normal values are <=2 lapses within the 10 minute test. Higher scores indicate worse vigilance.
Time Frame: Administered during diabetes education sessions done within the first 6 weeks of study; baseline, approximately 3 weeks after starting CPAP, and at the 2nd diabetes education session
Population: All randomized participants with data were were analyzed (the intention to treat method). This measure was not done per site protocol at West Virginia (n=12) and Detroit (n=1)), missing data from participants at Pittsburgh and VA Pittsburgh sites (n=29).
Measure: Mean (Standard Error); unit: transformed lapses
Arm/Group | Active CPAP Treatment | Sham-CPAP
Number analyzed (Participants) | 33 | 33
transformed lapses
  Baseline | 4.68 (0.45) | 4.67 (0.45)
  Average Lapses First Diabetes Session | 4.30 (0.47) | 3.56 (0.47)
  Average lapses 2nd Diabetes Education Session | 3.59 (0.54) | 4.78 (0.54)
Statistical Analysis 1: Comparison: Active CPAP Treatment vs Sham-CPAP; Test type: Superiority; p = 0.005, Mixed Models Analysis — F-test statistics for group X time = 5.66; Mean Difference (Net) = 0.006, 95% CI 2-sided [-1.27 to 1.28], Standard Error of Mean 0.64 — Treatment Difference = Active CPAP - Sham CPAP

ADVERSE EVENTS:
Time Frame: Until study completion, up to 36 weeks.
Description: Any adverse event was evaluated at the scheduled participant assessments at 6 weeks, 12 weeks, 24 weeks, and 36 weeks.
Groups:
- Active CPAP Following Sham-CPAP: Persons who completed 12-weeks on sham-CPAP, were debriefed, titrated for active CPAP
Arm/Group | Active CPAP Treatment | Sham-CPAP | Active CPAP Following Sham-CPAP
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/49 | 0/20
Serious Adverse Events (participants affected / at risk) | 1/49 | 1/49 | 0/20
Other Adverse Events (participants affected / at risk) | 0/49 | 2/49 | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active CPAP Treatment (N=49) | Sham-CPAP (N=49) | Active CPAP Following Sham-CPAP (N=20)
Infection in knees bilateral (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) — Hospitalization for 2 days for septic arthritis of knees bilaterally--unrelated to study.
Diagnosed with lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) — Unrelated to study but discharged from study
Hypertension (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) — Participant hospitalized for 2 days with hypertension.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active CPAP Treatment (N=49) | Sham-CPAP (N=49) | Active CPAP Following Sham-CPAP (N=20)
difficulty wearing mask (Product Issues) | 0 (0) | 2 (2) | 0 (0) — Complains of claustrophobia feelings while wearing the mask

LIMITATIONS AND CAVEATS:
Recruitment was negatively affected by a large number of persons screened who were ineligible because of either their, or a family member, having prior CPAP treatment. Recruitment was also affected by persons who did not want the possibility of being randomized to be on a sham-CPAP device for 12 weeks.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-12): https://cdn.clinicaltrials.gov/large-docs/55/NCT01901055/Prot_SAP_000.pdf